CLINICAL TRIAL: NCT06644144
Title: Early Identification of Progressive Pulmonary Fibrosis, Precision Medicine for More Oxygen - ILD Extension.
Brief Title: P4O2 ILD Extension
Acronym: P4O2-ILD
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: AbbVie (Industry); Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Jan Willem Duitman, Dr. Jan Willem Duitman, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2023.0591; NL84006.018.23 (Other: CCMO)
Record Dates: First submitted 2024-09-23; First posted 2024-10-16 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Interstitial Lung Disease; Pulmonary Fibrosis; Interstitial Lung Fibrosis; IPF; Pulmonary Fibrosis, Idiopathic; Pulmonary Fibrosis Idiopathic Familial; Chronic Hypersensitivity Pneumonitis; Unclassifiable ILD; Idiopathic NSIP; CTD-ILD
Keywords: Interstitial Lung Disease; Interstitial Lung Abnormalities; Progressive Pulmonary Fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, feces, breath analysis, nasal brush, Bronchoalveolar lavage fluid, lung biopsy, Particles in Exhaled Air (PExA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Idiopathic Pulmonary Fibrosis/Familial Pulmonary Fibrosis
  Interventions: Other: No Interventions
- fibrotic ILD: Patients with a diagnosis of: chronic Hypersensitivity Pneumonitis (cHP), unclassifiable ILD (uILD), idiopathic NSIP or CTD-ILD.
  Interventions: Other: No Interventions
- Interstitial Lung Abnormalities
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No intervention so not applicable.

SUMMARY:
The goal of this observational study is to identify early biomarkers that can predict the development of progressive pulmonary fibrosis (PPF) in participants with interstitial lung diseases (ILDs). The participant population includes adults diagnosed with idiopathic pulmonary fibrosis (IPF), familial pulmonary fibrosis (FPF), other fibrotic ILDs, and interstitial lung abnormalities (ILA).

The main questions it aims to answer are:

* What biomarkers and risk factors are linked to fibrosis progression or can predict rapid worsening and sudden flare-ups in IPF and FPF patients?
* What biomarkers and risk factors can predict the development of a PPF phenotype in different types of ILD?
* What biomarkers and risk factors can help identify ILA patients who may develop significant ILD?
* What biomarkers and risk factors can predict how well ILD patients will respond to treatment?

Researchers will compare the outcomes between participants diagnosed with IPF/FPF, other fibrotic ILDs, and ILA to see if early detection biomarkers differ among these groups.

Participants will:

* Undergo blood sampling.
* Perform lung function tests.
* Have CT scans.
* Perform breath analysis
* Participate in exposome and microbiome analyses.
* Complete questionnaires.
* A subgroup of participants will be offered bronchoscopy.

DETAILED DESCRIPTION:
Included participants will complete several study visits to collect clinical data and biological samples. Study visits will be performed at baseline, 3, 6, 12, 24, 36, 48 and 60 months, with a 2-month time window for follow-up visits. These time points are aligned with the standard clinical follow-up visits outlined in the ILD Care Path Protocol of Amsterdam UMC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of (1) idiopathic pulmonary fibrosis (IPF), familial pulmonary fibrosis (FPF), (2) other fibrotic ILDs (fILD), including fibrotic hypersensitivity pneumonitis (fHP), idiopathic non-specific interstitial pneumonia (iNSIP), connective tissue disease (CTD)-ILD, and unclassifiable ILD (uILD); or (3) interstitial lung abnormalities (ILA).
* Meeting all the following criteria during the screening period:

  1. FVC ≥45% predicted.
  2. FEV1/FVC ≥0.7.
  3. DLco corrected for Hb ≥40% predicted.
* Able to provide written informed consent as approved by the independent ethics committee.
* Able to undergo a CT scan and perform PFT.
* Age > 18 years and < 80 years.
* Understanding of the Dutch or English language.

Exclusion Criteria:

* Combined pulmonary fibrosis and emphysema (CPFE) diagnosis
* Chronic obstructive lung disease (COPD) with an FEV1/FVC <70%.
* Uncontrolled severe asthma.
* Active malignancy, except for squamous cell carcinoma of the skin, low-risk breast cancer, and low-risk prostate cancer.
* Pregnancy or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The P4O2 ILD-extension is a non-interventional prospective observational cohort study that will include a minimum of 450 participants, divided intro three groups (1) 150 participants diagnosed with idiopathic pulmonary fibrosis (IPF) or familial pulmonary fibrosis (FPF); (2) 150 participants diagnosed with other fibrotic ILDs (fILD), including fibrotic hypersensitivity pneumonitis (fHP), idiopathic non-specific interstitial pneumonia (iNSIP), connective tissue disease (CTD)-ILD, and unclassifiable ILD (uILD); and (3) 150 participants diagnosed with interstitial lung abnormalities (ILA).
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory and fibrosis extent assessed by HRCT | A baseline HRCT scan will be performed during screening. Following inclusion in the study, HRCT scans will be repeated annually, starting one year after the initial scan, and continuing each year until the end of follow-up (at 5 years))
  High-Resolution Computed Tomography (HRCT) is an advanced imaging technique used to obtain detailed images of the lungs and chest. Unlike standard CT scans, HRCT uses thin slices and special algorithms to produce high-resolution images that provide more precise visualization of lung structures, making it particularly useful for diagnosing and evaluating various lung conditions. The Inflammatory and Fibrosis extent will be analyzed by using artificial intelligence software.
Pulmonary function tests (PFTs)- Spirometry volumes | It will be measured at baseline, at 3, 6, and 12 months, and every other year till end of follow-up (60months))
  Pulmonary function tests (PFTs) are a group of tests that measure how well your lungs are working. These tests assess lung volume, capacity, rates of flow, and gas exchange. We will look at the following values:
  1. Spirometry Values
  * Forced Vital Capacity (FVC): The total amount of air exhaled after taking the deepest breath possible.
  * Forced Expiratory Volume in 1 Second (FEV1): The amount of air forcefully exhaled in one second.
Pulmonary function tests (PFTs)- DLCO measurement | It will be measured at baseline, at 3, 6, and 12 months, and every other year till end of follow-up (60months))
  Pulmonary function tests (PFTs) are a group of tests that measure how well your lungs are working. These tests assess lung volume, capacity, rates of flow, and gas exchange. We will look at the Diffusion Capacity Tests (DLCO). DLCO: Measures how well oxygen and CO2 are exchanged between the lungs and the blood.
Pulmonary function tests (PFTs)- Lungvolume measurement | It will be measured at baseline, at 3, 6, and 12 months, and every other year till end of follow-up (60months))
  Pulmonary function tests (PFTs) are a group of tests that measure how well your lungs are working. These tests assess lung volume, capacity, rates of flow, and gas exchange. We will look at the Lung Volumes and Capacities
  * Total Lung Capacity (TLC): The total volume of air in the lungs after taking the deepest breath.
  * Residual Volume (RV): The amount of air left in the lungs after a full exhalation.
  * Functional Residual Capacity (FRC): The amount of air remaining in the lungs after normal exhalation.
  * Inspiratory Capacity (IC): The maximum amount of air that can be inhaled after a normal exhalation.
Biomarkers related to pulmonary fibrosis will be measured in plasma and serum | It will be measured at baseline, at 3, 6, and 12 months, and every other year till end of follow-up (60months))
  Blood will be taken from participants at the 8 different time points. A predefined panel of biomarkers related to pulmonary fibrosis will be measured in serum/plasma, urine, and, if available, bronchoalveolar lavage fluid. Biomarker levels will be correlated with the time to event (i.e., development of rapid progression or acute exacerbation) to identify biomarkers that predict rapid progression or acute exacerbation, as defined by the criteria by Raghu et al., (2022).
Peripheral blood mononuclear cell (PBMC) populations in blood | It will be measured Will be measured at baseline, at 3, 6 months, 12 months, and every other year till end of follow-up (60months)
  Deep phenotyping of peripheral blood mononuclear cells (PBMCs) and, when available, BAL cells will be performed using flow cytometry, spectral flow, or cyTOF (cytometry by time of flight). A panel of surface and activation markers will define subsets of monocyte and lymphocyte populations. Data will be correlated to the time of the event.
Exhaled breath analysis including volatile organic compounds | It will be measured at baseline, at 3, 6, and 12 months, and every other year till end of follow-up (60months))
  Exhaled breath analysis involves measurements of volatile organic compounds (VOCs) using gas chromatography-mass spectrometry (GC-MS) and electronic sensor detection of exhaled breath compounds in a non-invasive manner (breathing into a device). For all participants, VOCs will be measured using GC-MS (in house GC mass spectrometer)..

SECONDARY OUTCOMES:
Disease-relevant questionnaires: Exposure Questionnaire | Questionnaires will be filled in at baseline, at 6, and 12 months, and every other year till end of follow-up (60months))
  During multiple visits, participants will be requested to complete the questionnaires below. The questionnaires that are not completed in the study center will be sent to the participants via email to fill out at home or bring to the clinic next visit. The Exposure questionnaire. Participants will be asked about their exposures and exposure risks. They are requested to answer the questions as completely as possible. The participant is asked about their current occupation and occupation history, as well as any present or past exposures to metals, fibers, chemicals, dust, smoke, fog/mist, gases, fumes, animal- or plant-materials, bacterial, viral or fungi contacts. Additionally, we will inquire about what kind of environment they have been living in and the duration of their residency. Other questions will cover hobbies, pesticide contact, and animal contact. The follow-up questionnaire has fewer questions.
Disease-relevant questionnaires: KBILD questionnaire. | Questionnaires will be filled in at baseline, at 6, and 12 months, and every other year till end of follow-up (60months))
  During multiple visits, participants will be requested to complete the questionnaires below. The questionnaires that are not completed in the study center will be sent to the participants via email to fill out at home. The King's Brief Interstitial Lung Disease (KBILD) questionnaire is designed to assess the impact of the ILD on the participant's overall well-being and daily life. It can be used to monitor the progression of ILD, evaluate treatment effectiveness, and assess ongoing management. The KBILD questionnaire consists of 15 brief items. For more details, please visit https://www.kbild.com.
Disease-relevant questionnaires: Modified Medical Research Council Dyspnea score | Questionnaires will be filled in at baseline, at 6, and 12 months, and every other year till end of follow-up (60months))
  During multiple visits, participants will be requested to complete the questionnaires below. The questionnaires that are not completed in the study center will be sent to the participants via email to fill out at home. The mMRC (Modified Medical Research Council) Dyspnea Scale is used to assess the level of baseline functional disability caused by dyspnea. The mMRC dyspnea scale ranges from grade 0 to 4, with 0 indicating minimal dyspnea. This longitudinal data is valuable for understanding the natural progression of ILDs and evaluating the effectiveness of long-term interventions.
Disease-relevant questionnaires: Visual analog scale (VAS) | Questionnaires will be filled in at baseline, at 6, and 12 months, and every other year till end of follow-up (60months))
  During multiple visits, participants will be requested to complete the questionnaires below. The questionnaires that are not completed in the study center will be sent to the participants via email to fill out at home. The Visual analog scale (VAS) is a linear scoring method with a scale ranging from 0 to 10. A score of 0 represents no coughing symptoms, while a score of 10 represents the most severe coughing. The participant is asked to mark the severity of the cough on the scale based on self-perception.
Disease-relevant questionnaires: Fatigue Severity Scale (FSS) | Questionnaires will be filled in at baseline, at 6, and 12 months, and every other year till end of follow-up (60months))
  During multiple visits, participants will be requested to complete the questionnaires below. The questionnaires that are not completed in the study center will be sent to the participants via email to fill out at home.
  The Fatigue Severity Scale (FSS) will be used to determine the severity of fatigue in participants. The questionnaire contains nine items and should take approximately 5 minutes to complete. Fatigue is assessed through nine statements that can be scored on a 7-point scale, ranging from 1 (strongly disagree) to 7 (strongly agree). The total score, ranging from 9 to 63, will be divided by 9. A higher score indicated a higher level of fatigue.
Genomics analysis in blood. | Genomics are done once at baseline.
  Increasing evidence suggests that genetic factors play a significant role in the emergence of interstitial lung disease (ILD), particularly within the framework of familial clustering, as seen in cases of familial interstitial pneumonia (FIP)(Borie et al., 2019).
  DNA and total RNA will be isolated from blood using the RNeasy DNA/RNA Universal kit (Qiagen). RNA will be used for generating the transcriptomic data, while DNA will be dedicated to GWAS analysis and methylome profiling. Whole genome transcriptome analysis will be conducted using state-of-the-art RNA sequencing.
Epigenomics analysis in blood. | Epigonomics are done at baseline and 1 year after inclusion.
  Increasing evidence suggests that genetic factors play a significant role in the emergence of interstitial lung disease (ILD), particularly within the framework of familial clustering, as seen in cases of familial interstitial pneumonia (FIP)(Borie et al., 2019).
  DNA and total RNA will be isolated from blood using the RNeasy DNA/RNA Universal kit (Qiagen). RNA will be used for generating the transcriptomic data, while DNA will be dedicated to GWAS analysis and methylome profiling. Whole genome transcriptome analysis will be conducted using state-of-the-art RNA sequencing.
Transcriptome analysis in blood. | Transcriptome is performed at baseline, 6 months and 1 year after inclusion.
  Increasing evidence suggests that genetic factors play a significant role in the emergence of interstitial lung disease (ILD), particularly within the framework of familial clustering, as seen in cases of familial interstitial pneumonia (FIP)(Borie et al., 2019).
  Whole genome transcriptome analysis will be conducted using state-of-the-art RNA sequencing. RNAseq libraries will be generated from poly-A enriched RNA and sequenced on the Illumina Hiseq sequencer. After sequencing, the generated reads will be aligned to the UCSC human hg19 reference genomes using software programs such as the short-read mappers and splice-junction identifier TopHat. Differential gene expression analysis will be performed using the DESeq package. RNAseq offers the advantage of detecting all expressed genes without any "a priori" selection through unlined microarray-based gene expression analysis.
Proteome analysis in bronchoalveolar lavage fluid | In Group 3, thirty participants will undergo bronchoalveolar lavage at baseline. Additional procedures may be performed during the follow-up period if clinically indicated and will be added to samples. .
  Biomarkerpanel related to pulmonary fibrosis will be measured in bronchoalveolar lavage fluid. A panel of biomarkers related to pulmonary fibrosis will be measured in BALF. The biomarkers will be determined using a biased approach using the Luminex® Instrument (Austin, USA) and unbiased approach using Olink® (Uppsala, Sweden) techniques. Units of Measure will be concentrations of the different proteins in picograms/mililiters
Microbiome analyses in stool and nasal swabs. | Once in first year
  The gut and respiratory microbiomes play an important role in regulating immune responses. The research study will assess the overall microbial metabolic activity and changes in microbiome composition by analyzing fecal and nasal samples from each participant.
Concentration of Biomarkers in Exhaled Particles (Collected via Impaction) | From moment of inclusion every year untill end of follow-up at 60 months.
  Small droplets, or particles, that arise when small airways close and re-open, are collected from the exhaled air and sampled by impaction (PExA technology). Biomarkers from exhaled air particles, collected through impaction, will be analyzed using proteomics platform assays or Enzyme-Linked Immunosorbent Assay (ELISA). The concentration of specific biomarkers (e.g., proteins, cytokines) will be quantified. Unit of Measure: Concentration (pg/mL or ng/mL).. For more details, visit https://pexa.se/en/.
Identification of Compounds in Exhaled Particles via Mass Spectrometry (MS) | From moment of inclusion every year untill end of follow-up at 60 months.
  Small droplets, or particles, that arise when small airways close and re-open, are collected from the exhaled air and sampled by impaction. Exhaled particles will be analyzed using Mass Spectrometry (MS) to identify and quantify specific compounds or molecular signatures. Concentration (μg/mL or relative abundance). For more details, visit https://pexa.se/en/.
Separation and Quantification of Compounds in Exhaled Particles Using Liquid Chromatography (LC) and High-Performance Liquid Chromatography (HPLC) | From moment of inclusion every year untill end of follow-up at 60 months.
  Small droplets, or particles, that arise when small airways close and re-open, are collected from the exhaled air and sampled by impaction. Liquid Chromatography (LC) and High-Performance Liquid Chromatography (HPLC) will be used to separate and quantify compounds present in exhaled air samples.
  Unit of Measure: Concentration (ng/mL or μg/mL). For more details, visit https://pexa.se/en/.
Metabolome analyses in blood. | Twice in the first year of inclusion; baseline and at 6 months.
  Metabolomics is a rapidly evolving field, and advancements in technology and analytical methods continue to enhance our understanding of the metabolome and its role in human health and disease. By profiling the metabolites present in blood, we can gain insights into metabolic pathways, identify disease signatures, monitor treatment response, and uncover potential therapeutic targets for ILD. IPF is associated with a distinct circulating metabolome (Hesslinger et al., 2019).
  Blood samples will be collected via venipuncture at ILD centers to profile metabolites associated with idiopathic pulmonary fibrosis (IPF). Specific biomarkers to be assessed include: Amino acids (e.g., glutamine, tryptophan), Lipids (e.g., triglycerides, phospholipids), Organic acids (e.g., lactate, citric acid), Nucleotides (e.g., ATP, uric acid). These metabolites will provide insights into metabolic pathways. Concentration (μmol/L, ng/mL, or similar, as appropriate for each metabolite).
Metabolome analyses in urine | Twice in the first year of inclusion; baseline and at 6 months.
  Metabolomics is a rapidly evolving field, and advancements in technology and analytical methods continue to enhance our understanding of the metabolome and its role in human health and disease. By profiling the metabolites present in blood, we can gain insights into metabolic pathways, identify disease signatures, monitor treatment response, and uncover potential therapeutic targets for ILD. IPF is associated with a distinct circulating metabolome (Hesslinger et al., 2019).
  Urine samples will be collected at home and stored at -80ºC in the biobank for metabolome and biomarker analysis. Specific biomarkers to be assessed include: Creatinine, Electrolytes (e.g., sodium, potassium), Organic metabolites (e.g., hippurate, citrate). These biomarkers will help identify metabolic changes related to ILD. Unit of Measure: Concentration (mmol/L, mg/mL, or similar, as appropriate for each metabolite).
Personal exposure to environmental pollutants using the Ultrasonic Personal Air Sampler | Exposome will be measured twice in first year, dependant on season (for most patients at 6 and 1 year follow-up))
  External exposome factors such as concentrations of ambient air pollution and other environmental pollutants will be quantified. Time-weighted measurements of PM2.5 will be collected using personal samplers.
External exposome analyses using Silicon wristbands | Exposome will be measured twice in first year, dependant on season (for most patients at 6 and 1 year follow-up))
  These wristbands collect exposome particles from the surrounding air in the participant's living environment. The wristbands will be worn for 4 to 5 days and then stored in a sealed bag to be returned to field workers. External exposome factors such as concentrations of ambient air pollution and other environmental pollutants will be quantified. Time-weighted measurements of PM2.5 will be collected.
External exposome analyses using a Sniffer-bike | Exposome will be measured twice in first year, dependant on season (for most patients at 6 and 1 year follow-up))
  Sniffer-bike will be placed at the home of the patient and measures external exposome factors such as concentrations of ambient air pollution and other environmental pollutants, these will be quantified. Time-weighted measurements of PM2.5 will be collected using these stationary samplers.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Nossent, MD, Principal Investigator — Amsterdam UMC, locatie VUmc; Jan Willem Duitman, PhD, Principal Investigator — Amsterdam UMC, locatie VUmc; Anke-Hilse Maitland-van der Zee, PhD, Principal Investigator — Amsterdam UMC, locatie VUmc
Locations (1):
- Amsterdam UMC, locatie VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The study is part of the P4O2 consortium, which focuses on chronic illnesses. Access to data is strictly regulated and provided only to answer research questions that emerge from an approved project proposal. The Data Committee evaluates whether a research question aligns with the original proposal and determines the specific conditions under which access is granted. Consortium members receive pseudonymized data for research and development purposes. These partners must sign a data sharing agreement before accessing the data. Private companies within the consortium may only receive anonymous data for commercial purposes. Private partners outside the consortium can request an analysis, but the outcome is limited to a report or scientific publication. For commercial purposes, these external private companies are permitted to receive only pseudonymized data, ensuring strict adherence to data protection protocols and ethical standards.